CLINICAL TRIAL: NCT02319070
Title: Prospective, Observational, 2-cohort Study of Adult Patients With Severe Hemophilia A in Greece. Cost,Clinical Outcomes and Quality of Life Comparison Between on Demand and Secondary Prophylaxis Treatment Strategies
Brief Title: 2-cohort Study of Adult Patients With Severe Hemophilia A in Greece
Acronym: HAMLET
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17493; KG1411GR (Other: Company Internal)
Record Dates: First submitted 2014-12-12; First posted 2014-12-18 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Hemophilia A
Keywords: Cost; Clinical Outcomes; Quality of Life; On Demand Treatment; Secondary Prophylaxis
MeSH Terms: conditions — Hemophilia A | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Adult patients with severe Hemophilia A.(25 patients on Secondary Prophylaxis treatment)
  Interventions: Other: Survey
- Cohort 2: Adult patients with severe Hemophilia A.(50 patients on On Demand treatment)
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Recombinant antihemophilic factor VIII (FVIII) on Secondary Prophylaxis treatment scheduled according to daily routine
  Groups: Cohort 1
Other: Survey — Recombinant antihemophilic factor VIII (FVIII) On Demand treatment scheduled according to daily routine
  Groups: Cohort 2

SUMMARY:
This study is a prospective, single center, observational, 2-cohort study of adult patients with severe Hemophilia A. There is no randomization procedure and all patients will be treated as per usual clinical practice. Patients will be followed up for 18 months after enrolment.

DETAILED DESCRIPTION:
The primary therapy for hemophilia is coagulation factor replacement, given either episodically on demand (OD) for the treatment of acute bleeds or prophylactically to prevent them.

The last years there has been an interest to study the comparative effectiveness of OD vs. SP (Secondary Prophylaxis) treatment strategies so as to create an evidence based platform to guide both clinical decision making and quantify the economic aspects of each treatment alternative. In Greece relevant information is lacking, thus it is imperative to study how patients on different treatment strategies are managed in a real-life setting in Greece, including the main factors associated with increased health care utilization, clinical success and patient well being.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe Hemophilia A.
* Age ≥18 years old
* Patients able to read and write
* Patients receiving Factor VIII substitute therapy, either on-demand or as secondary prophylaxis.
* Patients under the same therapeutic strategy (On Demand or Secondary Prophylaxis) for at least 6 months prior to enrolment.

Exclusion Criteria:

* Patients that have developed inhibitors against factor VIII.
* Patients participating in an investigational program with interventions outside of routine clinical practice.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a single center prospective two-cohort observational study conducted in a hospital setting.Patients will be enrolled from the biggest specialty management center in Greece
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Annual direct medical cost of specialized hemophilia centre for patients with the on-demand strategy | At 18 months
Annual direct medical cost of specialized hemophilia centre for patients with secondary prophylaxis | At 18 months

SECONDARY OUTCOMES:
Mean cost per joint bleed episodes for overall patients | At 18 months
Mean cost per joint bleed episodes by cohort for patients | At 18 months
Number of joint bleed episodes for overall patients | At 18 months
Number of joint bleed episodes by cohort for patients. | At 18 months
Severity of joint bleed episodes for overall patients. | At 18 months
Severity of joint bleed episodes by cohort for patients. | At 18 months
Mean EQ-VAS score as reported from patients at the time of a major bleed. | At 18 months
  EQ-VAS score is Standardized questionnaire for hemophilia
Mean EQ-5D score as reported from patients at the time of a major bleed. | At 18 months
  EQ-5D The EuroQol standardized instrument of health outcome
Mean change from baseline in Quality of Life scores derived from the Haem-A-Qol and EQ-5D questionnaires | Baseline and at 18 months
  Haem-A-Qol Specific questionnaire for hemophilia and EQ-5D The EuroQol standardized instrument of health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Greece